CLINICAL TRIAL: NCT00002866
Title: A Phase I/II Study of Docetaxel and Epirubicin as First-Line Therapy for Metastatic Breast Cancer
Brief Title: Docetaxel and Epirubicin With and Without G-CSF in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Purpose: Treatment
Other Study IDs: MA15; CAN-NCIC-MA15; NCI-V96-1063; CDR0000065138 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Neutropenia
Keywords: stage IV breast cancer; recurrent breast cancer; neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — Filgrastim; Docetaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: filgrastim
Drug: docetaxel
Drug: epirubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as G-CSF may increase the number of immune cells found in bone marrow or peripheral blood and may help a person 's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of docetaxel and epirubicin with and without G-CSF in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and recommended phase II dose of docetaxel in combination with epirubicin and filgrastim (G-CSF) as first-line therapy in women with metastatic breast cancer (phase II closed as of 03/27/2000). II. Determine the pharmacokinetic profile of docetaxel and epirubicin in these patients. III. Evaluate the toxicity of this regimen given at the recommended phase II dose. IV. Determine the response rate and duration of response in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of epirubicin and docetaxel. Patients receive epirubicin IV over 15 minutes followed by docetaxel IV over 60 minutes on day 1. Patients also receive filgrastim (G-CSF) subcutaneously on days 4-13. Treatment continues every 3 weeks for at least 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of epirubicin and docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose in which at least 2 of 6 patients experience dose-limiting toxicity. Additional patients will be accrued to receive treatment at the recommended phase II dose (phase II closed as of 03/27/2000). Patients are followed at 1 month and then every 3 months for survival.

PROJECTED ACCRUAL: Approximately 15-20 patients will be accrued within 4-5 months for the phase I portion of the study. A total of 15-30 patients will be accrued within 7-8 months for the phase II portion of the study (closed as of 03/27/2000).

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed breast cancer Newly diagnosed or progressive metastatic disease with at least 1 metastatic target lesion No known clinical brain or leptomeningeal metastasis Phase I entry: Measurable and/or evaluable disease with an indicator lesion outside prior radiotherapy field Phase II entry: (closed as of 03/27/2000) Bidimensionally measurable disease with an indicator lesion outside prior radiotherapy field At least 1 x 1 cm on chest x-ray At least 2 x 2 cm on CT scan or ultrasound Skin lesion or node at least 1 x 1 cm No bone-only lesion Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 16 and over Sex: Female Menopausal status: Not specified Performance status: ECOG 0-2 Hematopoietic: Absolute granulocyte count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than the upper limit of normal (ULN) AST/ALT no greater than 1.5 times ULN Alkaline phosphatase no greater than 2.5 times ULN (no greater than 5.0 times ULN if AST/ALT normal) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: Left ventricular ejection fraction at least 50% at rest by MUGA or echocardiogram No congestive heart failure No angina pectoris (even if controlled) No myocardial infarction within the past year No uncontrolled arrhythmia No uncontrolled hypertension Other: No active infection No grade 2 or greater symptomatic peripheral neuropathy No significant neurologic or psychiatric disorder, including dementia or seizures No peptic ulcer, unstable diabetes mellitus, or other contraindication to dexamethasone No prior malignancy except nonmelanomatous skin cancer or excised carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception Geographically accessible

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent supportive colony-stimulating factors (e.g., filgrastim (G -CSF)) (Prophylactic treatment during the second step of phase I allowed) Chemotherapy: Phase I patients: At least 12 months since prior adjuvant chemotherapy Prior neoadjuvant chemotherapy allowed Prior cumulative dose of doxorubicin no greater than 300 mg/m2 Prior cumulative dose of epirubicin no greater than 500 mg/m2 If epirubicin dose level at least 90 mg/m2: Prior cumulative dose of doxorubicin no greater than 200 mg/m2 Prior cumulative dose of epirubicin no greater than 300 mg/m2 Phase II patients: (closed as of 03/27/2000) No prior neoadjuvant or adjuvant chemotherapy regimen other than cyclophosphamide, methotrexate, and fluorouracil, or doxorubicin and cyclophosphamide given for a maximum of 4 courses All patients: No prior chemotherapy for metastatic disease No prior taxanes Endocrine therapy: Prior hormonal therapy in the adjuvant and/or metastatic setting allowed if subsequent disease progression No more than 2 prior hormonal therapy regimens for metastatic disease No concurrent corticosteroids (except for premedication or hypersensitivity reaction) Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy (unless single fractions for palliation) Concurrent local palliative radiotherapy for control of bone pain or for other reasons with no curative intent allowed Concurrent whole-brain radiotherapy for brain metastasis allowed No concurrent radiotherapy to sole measurable lesion Surgery: Not specified Other: No other concurrent investigational drugs or anticancer therapy No concurrent preventive IV antibiotics

Ages: 16 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1996-08-12 (Actual); Primary Completion 2005-07-19 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E. Trudeau, BSc, MA, MD, FRCPC, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (6):
- Canada (6):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Women's College Campus, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Hotel Dieu de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No